CLINICAL TRIAL: NCT00001505
Title: The Acquisition of Blood and Skin Samples From Patient Volunteers to Support Research Activities on Dermatologic and Other Diseases
Brief Title: The Acquisition of Blood and Skin Samples From Normal Volunteers to Support Research Activities on Dermatologic Diseases
Status: Completed | Type: Observational
Sponsor: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960097; 96-AR-0097
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2026-02-05 (Actual); Status verified 2026-01-22

CONDITIONS: Healthy Volunteer; Dermatologic Diseases; Systemic Diseases
Keywords: Biopsy; Research; Autoimmune; Blistering; Compensation; Natural History
MeSH Terms: conditions — Skin Diseases; Blister

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1/Single Cohort: Healthy individuals (including employees and other patients) and patients with selected skin or other diseases

SUMMARY:
Background:

-This protocol is concerned with the acquisition of blood, skin, or mucosal samples from healthy volunteers or patients with selected skin diseases to support the basic science and clinical research activities of the Dermatology Branch and other intramural Laboratories and Branches at the NIH Clinical Research Center.

Objectives:

(Primary)

-To allow collection of blood, skin, or mucosal samples from healthy volunteers or patients with selected skin or systemic diseases as needed to support the research activities of our Branch and other Laboratories and Branches.

Eligibility:

* Healthy individuals (including employees and other patients) and patients with selected skin or other diseases, including individuals of both genders and all racial/ethnic groups.
* Patient volunteers must be willing to undergo blood drawing and/or skin/mucosal biopsies.

Design:

-This is dependent upon the particular investigation for which these samples are needed....

DETAILED DESCRIPTION:
Background:

-This protocol is concerned with the acquisition of blood, skin, or mucosal samples from healthy volunteers or patients with selected skin diseases to support the basic science and clinical research activities of the Dermatology Branch and other intramural Laboratories and Branches at the NIH Clinical Research Center.

Objectives:

(Primary)

-To allow collection of blood, skin, or mucosal samples from healthy volunteers or patients with selected skin or systemic diseases as needed to support the research activities of our Branch and other Laboratories and Branches.

Eligibility:

* Healthy individuals (including employees and other patients) and patients with selected skin or other diseases, including individuals of both genders and all racial/ethnic groups.
* Patient volunteers must be willing to undergo blood drawing and/or skin/mucosal samples/monitoring.

Design:

-This is dependent upon the particular investigation for which these samples are needed.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy individuals (including employees and other patients), and patients with selected skin or other diseases, including individuals of both genders and all racial/ethnic groups.

Patient volunteers must be willing to undergo blood drawing and/or skin/mucosal sampling/monitoring to include non-invasive skin samples.

EXCLUSION CRITERIA:

Strong family history and/or evidence of keloid formation following surgery or trauma.

Children under the age of 18 years.

Pregnant women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers or patients with selected skin diseases
Sampling Method: Non-Probability Sample
Enrollment: 304 (Actual)
Dates: Start 1998-01-15 (Actual)

PRIMARY OUTCOMES:
Collection of blood, skin, or mucosal samples from healthy volunteers or patients with selected skin or systemic diseases | Ongoing
  Collection of blood, skin, or mucosal samples from healthy volunteers or patients with selected skin or systemic diseases

CONTACTS AND LOCATIONS:
Overall Officials: Heidi H Kong, M.D., Principal Investigator — National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1996-AR-0097.html